CLINICAL TRIAL: NCT02186990
Title: Comparison of Etomidate, Propofol and Etomidate-propofol Combination in Terms of Effects on Haemodynamic Response to Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, özgür yağan, MD, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Odu-2
Record Dates: First submitted 2014-06-06; First posted 2014-07-10 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Induction of Anaesthesia
MeSH Terms: interventions — Propofol; Etomidate

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- propofol (Active Comparator)
  Interventions: Drug: etomidate-propofol
- etomidate (Active Comparator)
  Interventions: Drug: etomidate
- propofol-etomidate (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — 2,5 mg/kg
  Arms: propofol-etomidate
Drug: etomidate — 0,3 mg/kg
  Arms: etomidate
Drug: etomidate-propofol — 0,15 mg/kg etomidate + 1,25 mg/kg propofol
  Arms: propofol

SUMMARY:
The purpose of this study is to evaluate the effect of propofol, etomidate and propofol-etomidate combination on hemodynamic responses during laryngoscopy and tracheal intubation and assess the adverse effect related to this drugs.

ELIGIBILITY:
Inclusion Criteria:

* between 18 - 65 age
* ASA I - II status
* elective surgery

Exclusion Criteria:

* emergency surgery
* pregnancy
* alcohol and drug abuse
* HT and cardiovascular disease
* BMI > 25 kg/m2
* hypersensitivity against study drug
* sedative drug use in last month
* difficult intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
haemodynamic values | in ten minutes after intubation
  e.g., heart rate, blood pressure (mean arterial pressure)

SECONDARY OUTCOMES:
adverse effect of study drugs | within in 30 minutes drug administration
  e.g. myoclonus, injection pain, allergy, skin rash

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Reanimation Dept. Ordu University Training and Research Hospital, Altinordu, Ordu, Turkey (Türkiye)